CLINICAL TRIAL: NCT05104476
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multi-centre Study to Assess the Efficacy, Safety and Tolerability of Lu AF82422 in Patients With Multiple System Atrophy
Brief Title: A Study of Lu AF82422 in Participants With Multiple System Atrophy
Acronym: AMULET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18331A
Record Dates: First submitted 2021-10-15; First posted 2021-11-03 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; Neurodegenerative Disorder; Autonomic Failure
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases; Pure Autonomic Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lu AF82422 (Experimental): Participants in the DBP will receive Lu AF82422 intravenous (IV) infusion every 4 weeks (Q4W) from Baseline for a minimum 48 weeks up to a maximum 72 weeks. In the optional OLE, all participants will receive Lu AF82422 IV infusion starting on Day 1 of the OLE up to week 188.
  Interventions: Drug: Lu AF82422
- Placebo (Experimental): Participants in the DBP will receive Lu AF82422 matching placebo IV infusion Q4W from Baseline for a minimum 48 weeks up to a maximum 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AF82422 — Solution for infusion
  Arms: Lu AF82422
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
To find out the effect of Lu AF82422 on disease progression in participants with multiple system atrophy.

DETAILED DESCRIPTION:
This study will consist of a double-blind period (DBP) and will include an optional open-label treatment extension (OLE) period. Participants in the DBP will be randomized to Lu AF82422 or placebo (2:1). All participants entering the OLE will receive Lu AF82422 during the OLE.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant is diagnosed with possible or probable MSA of the multiple system atrophy parkinsonian type (MSA-P) or multiple system atrophy cerebellar type (MSA-C) sub-type at the Screening Visit.
* The participant had onset of motor and/or autonomic (orthostatic or urinary) MSA symptoms within 5 years prior to the Screening Visit in the judgement of the investigator.
* The participant has an UMSARS Part I score ≤16 (omitting item 11 on sexual function) at the Screening Visit.
* The participant has a cognitive performance evaluated by the Montreal Cognitive Assessment (MoCA) with a score ≥22 at the Screening Visit.

Open-label Extension Entry Criteria

* The participant has completed the EoT Visit and did not withdraw in the DBP.
* The participant has consented to participate in the OLE.
* The participant has completed the DBP within the last 5 months and will be enrolled into the OLE no later than end of Q1 2024.
* The participant is, in the Investigator's opinion, likely to comply with the protocol.
* The participant has not received any other Investigational product since the EOoTDBP Visit.

Key Exclusion Criteria:

* The participant has been treated with an anti-α-synuclein monoclonal antibody, mesenchymal stem cells or an inhibitor of α-synuclein aggregation within the last 12 months.
* The participant has any past or current treatment with an active vaccine targeting α-synuclein.
* The participant has 2 or more blood relatives with a history of MSA.
* The participant has evidence (clinically or on MRI) and/or history of any clinically significant disease or condition other than MSA (for example, serious neurological disorder, other intracranial disease, or systemic disease).
* The participant has a current diagnosis of movement disorders that could mimic MSA (for example, Parkinson' disease, dementia with Lewy bodies, essential tremor, progressive supranuclear palsy, spinocerebellar ataxia, spastic paraparesis, corticobasal degeneration, or vascular, pharmacological, or post-encephalitic parkinsonism), per investigator discretion.

Other inclusion and exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2028-03-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (19):
- United States (16):
  - The Parkinsons and Movement Disorder Institute, Fountain Valley, California
  - University of California - San Diego, La Jolla, California
  - University of California, San Francisco Neurosciences Clinical Research Unit, San Francisco, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Parkinson's Disease And Movement Disorder Center Of Boca Raton, Boca Raton, Florida
  - University of Florida Norman Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Rush University Medical Center, Rush University Cancer Center, Chicago, Illinois
  - Endeavor Health - Glenbrook Hospital, Glenview, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Health Medical Center, New York, New York
  - Columbia University Medical Center - The Neurological Institute of New York, New York, New York
  - Penn State Milton S. Hershey Medical Center - Penn State Hershey Neuroscience Institute (PSHNI), Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
- Japan (3):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Gifu University Hospital, Gifu, Gifu
  - National Hospital Organization Sendai Nishitaga Hospital, Sendai, Miyagi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a Placebo-controlled Double-blind Period (DBP) (48 weeks up to 72 weeks) and an Optional Open-label Extension (OLE) Period (96 weeks). Individual participant End of Trial (EOT) DBP will vary from 48 to 72 weeks. Once the last participant reaches week 48, the remaining participants will have their next scheduled visit converted to EOT DBP.
Pre-assignment Details: The data for DBP has been reported. The optional OLE period data will be reported after study completion.
Groups:
- Placebo: Participants received Lu AF82422 matching placebo IV infusion Q4W from Baseline for a minimum 48 weeks up to a maximum 72 weeks in the DB period.
- Lu AF82422: Participants received Lu AF82422 IV infusion Q4W from Baseline for a minimum 48 weeks up to a maximum 72 weeks in the DB period.
Period: Overall Study
Arm/Group | Placebo | Lu AF82422
Started | 22 | 42
Received at Least 1 Dose of Study Drug | 21 | 40
Completed | 16 | 32
Not Completed | 6 | 10
Not completed — Randomized But Not Treated | 1 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other Than Specified | 0 | 3

BASELINE CHARACTERISTICS:
Population: All-patients-treated set (APTS) included all randomized participants who took at least 1 dose of double-blind investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lu AF82422 | Total
Number analyzed (Participants) | 21 | 40 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (6.85) | 61.4 (8.09) | 60.8 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 11 | 21 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 12 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 26 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Unified Multiple System Atrophy Rating Scale (UMSARS) Part I and Part II Total Score (UMSARS TS) [Mean (Standard Deviation); unit: units on a scale] — UMSARS TS was obtained by sum of items from Part I and Part II. Part I assesses historical information on symptoms and activities of daily living (12 items) rated on a scale ranging from 0 (not affected) to 4 (unable to do activity). Part I total score range: 0 to 48. Part II consists of a clinical examination of key multiple system atrophy (MSA) motor signs and symptoms (14 items) rated on a scale ranging from 0 (normal) to 4 (severe impairment). Part II total score range: 0 to 56. UMSARS TS ranged from 0 (no impairment) to 104 (severe impairment). A higher score indicated greater impairment.
  units on a scale | 37 (7.77) | 34.8 (9) | 35.5 (8.59)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Slowing of Clinical Progression Based on Change From Baseline in the UMSARS TS at the End of Treatment (EOT) DB Period (DBP)
Description: The primary endpoint assessed disease progression by a Bayesian repeated measures model on UMSARS TS. Reported here is the estimated slowing (%) of clinical progression in participants receiving Lu AF82422 relative to those receiving placebo. UMSARS is a combined clinician and patient-reported outcome assessment developed to provide a surrogate measure of disease progression in multiple system atrophy (MSA). UMSARS TS was obtained by the sum of the items from Part I and Part II. Part I assesses historical information on symptoms and activities of daily living over the past 2 weeks and Part II consists of a clinical examination of key MSA motor signs and symptoms. UMSARS TS score was the sum of all items and ranged from 0 (no impairment) to 104 (severe impairment). A higher score indicated greater impairment.
Time Frame: Baseline up to Week 72
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of double-blind IMP and had a valid baseline assessment and at least 1 valid post-baseline assessment of the UMSARS TS, prior to, or at withdrawal from treatment.
Measure: Number; unit: Percentage Slowing of Clin. Progression
Groups:
- Lu AF82422 or Placebo: Participants received Lu AF82422 or Placebo IV infusion Q4W from Baseline for a minimum of 48 weeks up to a maximum 72 weeks in the DB period.
Arm/Group | Lu AF82422 or Placebo
Number analyzed (Participants) | 61
Percentage Slowing of Clin. Progression | 19
Statistical Analysis 1: Comparison: Lu AF82422 or Placebo; Test type: Superiority; Bayesian Progression Model = 0.81, 95% CI 2-sided [0.56 to 1.13] — Reported here is the estimated effect parameter from the Bayesian Progression Model and the associated Credibility Interval for the active arm

2. Secondary Outcome: Change From Baseline in the UMSARS TS at the End of Treatment (EOT) DBP
Description: UMSARS is a combined clinician and patient-reported scale to assess motor impairment in MSA participants. UMSARS TS was obtained by the sum of the items from Part I and Part II. Part I assesses historical information on symptoms and activities of daily living over the past 2 weeks (12 items) rated on a scale ranging from 0 = not affected to 4 = unable to do the activity. Part I total score ranged between 0 to 48 (higher score indicated greater impairment). Part II consists of a clinical examination of key MSA motor signs and symptoms (14 items) rated on a scale ranging from 0 = normal to 4 = marked/severe impairment. Part II total score ranged between 0 and 56 (higher score indicated greater impairment). UMSARS TS score was the sum of all 26 items and ranged from 0 (no impairment) to 104 (severe impairment). A higher score indicated greater impairment. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Weeks 48 and 72
Population: FAS included all randomized participants who received at least 1 dose of double-blind IMP and had a valid baseline assessment and at least 1 valid post-baseline assessment of the UMSARS TS, prior to, or at withdrawal from treatment. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 37
units on a scale
  Change at Week 48 | 13.93 (3.42) | 13.32 (2.86)
  Change at Week 72: number analyzed (Participants) | 5 | 14
  Change at Week 72 | 19.13 (3.74) | 15.10 (3.00)

3. Secondary Outcome: Change From Baseline in the Modified UMSARS Part I (mUMSARS) Score at the EOT DBP
Description: UMSARS Part 1 assesses historical information on symptoms and activities of daily living over the past 2 weeks as reported by participants and caregivers (12 items) rated on a scale ranging from 0 to 4; with 0 = not affected/normal 1= mildly affected/impaired, 2= moderately affected/impaired, 3= severely affected/impaired, and 4 = helpless or entirely affected/impaired. The modified UMSARS part I (mUMSARS) score was derived by collapsing the response option 0 and 1 within each item (0 & 1 =1). Hence, the mUMSARS score ranged from 12 to 48 (higher score indicated greater impairment). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Weeks 48 and 72
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 17 | 38
units on a scale
  Change at Week 48 | 7.07 (1.62) | 6.48 (1.33)
  Change at Week 72: number analyzed (Participants) | 5 | 15
  Change at Week 72 | 8.40 (2.00) | 8.77 (1.44)

4. Secondary Outcome: Change From Baseline in the UMSARS Part I Scores at the EOT DBP
Description: UMSARS Part 1 assesses historical information on symptoms and activities of daily living over the past 2 weeks as reported by participants and caregivers (12 items: speech, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, walking, falling, orthostatic symptoms, urinary function, sexual function, and bowel function) each rated on a scale ranging from 0 to 4; with 0 = not affected/normal 1= mildly affected/impaired, 2= moderately affected/impaired, 3= severely affected/impaired, and 4 = helpless or entirely affected/impaired. Part I total score ranged between 0 to 48 (higher score indicated greater impairment). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Weeks 48 and 72
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 17 | 38
units on a scale
  Change at Week 48 | 7.64 (1.92) | 6.98 (1.59)
  Change at Week 72: number analyzed (Participants) | 5 | 15
  Change at Week 72 | 8.49 (2.21) | 10.23 (1.65)

5. Secondary Outcome: Change From Baseline in the UMSARS Part II Scores at the EOT DBP
Description: UMSARS Part II consists of a clinical examination of key MSA motor signs and symptoms (14 items: facial expression, speech, ocular motor dysfunction, tremor at rest, action tremor, increased tone, rapid alternating movements of hands, finger taps, leg agility, heel-knee-shin test, arising from chair, posture, body sway, gait) each rated on a scale ranging from 0 to 4; with 0 = not affected/normal 1= mildly affected/impaired, 2= moderately affected/impaired, 3= severely affected/impaired, and 4 = helpless or entirely affected/impaired. Part II total score ranged between 0 and 56 (higher score indicated greater impairment). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Weeks 48 and 72
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 37
units on a scale
  Change at Week 48 | 7.16 (2.15) | 6.76 (1.83)
  Change at Week 72: number analyzed (Participants) | 5 | 14
  Change at Week 72 | 10.24 (2.38) | 7.10 (1.93)

6. Secondary Outcome: Change From Baseline in Schwab and England Activities of Daily Living (SE-ADL) Score at Week 48 in the DBP
Description: The SE-ADL is a combined participant- and clinician-reported scale to assess participants physical functioning in activities in daily living to grade functional status. For this study, only the clinician-rated part was administered. The SE-ADL scale uses percentages to represent how much effort and dependence on others, participants need to complete daily chores. The SE-ADL scale ranged from 0% indicating worst possible function (fully dependent) to 100% indicating no impairment (completely independent). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: FAS included all randomized participants who received at least 1 dose of double-blind IMP and had a valid baseline assessment and at least 1 valid post-baseline assessment of the UMSARS TS, prior to, or at withdrawal from treatment. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 36
units on a scale | -23.56 (7.40) | -20.82 (6.52)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score at Week 48 in the DBP
Description: The CGI-S was administered by an experienced neurologist familiar with MSA participants to make an expert clinical global judgement about the severity of the disease across various time points. The rating was based upon observed and reported symptoms, behaviour, and function in the past seven days. The CGI-S was rated on a scale ranging from 0 to 4 (whereas the 0 = normal, not impaired; 1 = mildly impaired; 2 = moderately impaired; 3 = severely impaired; 4 = extremely impaired). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 36
units on a scale | 0.58 (0.17) | 0.34 (0.14)

8. Secondary Outcome: Change From Baseline in Patient Global Impression - Severity of Illness (PGI-S) Score at Week 48 in the DBP
Description: The PGI-S is a self-reported single item to evaluate all aspects of participants' MSA symptoms. Participants were asked to choose the response that best described the severity of their MSA symptoms over the past week. The question was rated on a 5-point scale ranging from 0 to 4 (0 = none; 1 = minor; 2 = moderate; 3 = severe; 4 = very severe). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 36
units on a scale | -0.07 (0.21) | 0.18 (0.18)

9. Secondary Outcome: Change From Baseline in Observer-Reported Global Impression - Severity of Illness (OGI-S) Score at Week 48 in the DBP
Description: The OGI-S is a single-question carer/observer-reported outcome to evaluate all aspects of participants' MSA symptoms. Carer/observers were asked to choose the response that best described the observed severity of MSA symptoms in the person they care for over the past week. The question was rated on a 5-point scale ranging from 0 to 4 (0 = none; 1 = minor; 2 = moderate; 3 = severe; 4 = very severe). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 11 | 16
units on a scale | 0.36 (0.22) | 0.20 (0.18)

10. Secondary Outcome: Composite Autonomic Symptom Score Select Change (COMPASS Select Change) Total Score at Week 48 in the DBP
Description: The COMPASS Select, a participant-reported scale, consists of a subset of 36 items derived from the original COMPASS, to assess severity of autonomic symptoms in MSA during the last year. The COMPASS Select includes 3 domains related to blood pressure control: syncope, orthostatic intolerance, and vasomotor symptoms; and 3 domains focused on symptoms of disturbed secretomotor, bladder, and sleep function. The COMPASS Select Change is a derivate of COMPASS Select, consisting of 16 items in which participants were asked to score their change in autonomic symptoms since their last visit. The scoring algorithm of COMPASS was highly complicated and required computer analysis for score generation. COMPASS Change Select score ranged from -150 to 150. A higher score indicated greater autonomic symptom severity.
Time Frame: Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 17 | 38
units on a scale | 18.79 (41.98) | 34.28 (26.86)

11. Secondary Outcome: Change From Baseline in UMSARS Part IV Score at Week 48 in the DBP
Description: The UMSARS part IV comprised a global disability scale ranging from 1-5, with 1 = 'Completely independent. Able to do all chores with minimal difficulty or impairment. Essentially normal. Unaware of any difficulty'; 2 = 'Not completely independent. Needs help with some chores'; 3 = 'More dependent. Help with half of chores. Spends a large part of the day with chores'; 4 = 'Very dependent. Now and then does a few chores alone or begins alone. Much help needed'; and 5 = 'Totally dependent and helpless. Bedridden'. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 17 | 38
units on a scale | 1.35 (0.35) | 1.13 (0.30)

12. Secondary Outcome: Change From Baseline in Speech, Swallowing, Falls, and Walking, as Assessed by the UMSARS Part I Item Scores at Week 48 in the DBP
Description: UMSARS Part I assesses historical information on symptoms and activities of daily living over the past 2 weeks as reported by participants and caregivers (12 items: speech, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, walking, falling, orthostatic symptoms, urinary function, sexual function, and bowel function) each rated on a scale ranging from 0 to 4; with 0 = not affected/normal 1= mildly affected/impaired, 2= moderately affected/impaired, 3= severely affected/impaired, and 4 = helpless or entirely affected/impaired. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 17 | 38
units on a scale
  Speech | 0.61 (0.26) | 0.19 (0.21)
  Swallowing | 0.57 (0.30) | 0.91 (0.25)
  Falls | 0.36 (0.42) | 0.22 (0.36)
  Walking | 1.02 (0.27) | 0.86 (0.23)

13. Secondary Outcome: Change From Baseline in Number of Falls, as Assessed by the Fall Diary Periods (Weeks 44 to 48) in the DBP
Description: Fall Diary period was defined as the period between the two visits where the diary was filled out according to the protocol. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Weeks 44 to 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: falls
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 15 | 33
falls | -0.18 (0.05) | -0.16 (0.04)

14. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension, 5-Level (EQ-5D-5L) Score at Week 48 in the DBP
Description: The EQ-5D-5L is a participant-reported assessment designed to measure the participant's wellbeing. It consisted of 5 descriptive items (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and a visual analogue scale (VAS) of the overall health state. Each descriptive item was rated on a 5-point index ranging from 1 (no problems) to 5 (extreme problems). The VAS ranged from 0 (worst imaginable health state) to 100 (best imaginable health state). LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 35
units on a scale
  Mobility Score | 0.75 (0.32) | 0.49 (0.28)
  Self Care Score | 0.80 (0.38) | 0.74 (0.32)
  Usual Activities Score | 0.50 (0.39) | 0.87 (0.34)
  Pain/Discomfort Score | -0.06 (0.38) | 0.22 (0.33)
  Anxiety/Depression Score | 0.05 (0.29) | 0.34 (0.25)
  VAS Score | -13.16 (6.46) | -13.80 (5.74)

15. Secondary Outcome: Percent Change From Baseline in Brain Volume With Ventricles, as Measured by Volumetric MRI (vMRI) at Week 48 in the DBP
Description: LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 37
percent change | -1.14 (0.39) | -0.81 (0.33)

16. Secondary Outcome: Percent Change From Baseline in P-Neurofilament Light Chain (NfL) Protein Concentration at Week 48 in the DBP
Description: LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lu AF82422
Number analyzed (Participants) | 16 | 36
percent change | 10.37 (11.60) | 6.81 (10.01)

17. Secondary Outcome: Lu AF82422 Plasma Concentration in the DBP
Time Frame: Weeks 0, 4, 6, 8, 12, 24, 36, 48, 60, 72, 88
Population: APTS included all randomized participants who received at least 1 dose of double-blind IMP. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Lu AF82422
Number analyzed (Participants) | 40
nanograms (ng)/milliliter (mL)
  Week 0 | NA (NA) — All observations at Week 0 were below the lower limit of quantification
  Week 4: number analyzed (Participants) | 37
  Week 4 | 186754 (63989)
  Week 6: number analyzed (Participants) | 34
  Week 6 | 408806 (148195)
  Week 8: number analyzed (Participants) | 38
  Week 8 | 285079 (170320)
  Week 12: number analyzed (Participants) | 39
  Week 12 | 312451 (128006)
  Week 24: number analyzed (Participants) | 39
  Week 24 | 418385 (349787)
  Week 36: number analyzed (Participants) | 38
  Week 36 | 417758 (170012)
  Week 48: number analyzed (Participants) | 36
  Week 48 | 390751 (181489)
  Week 60: number analyzed (Participants) | 33
  Week 60 | 526706 (312743)
  Week 72: number analyzed (Participants) | 14
  Week 72 | 544071 (355696)
  Safety Follow Up (Week 88): number analyzed (Participants) | 4
  Safety Follow Up (Week 88) | 42425 (18372)

18. Secondary Outcome: Lu AF82422 Cerebrospinal Fluid (CSF) Concentrations in the DBP
Time Frame: Weeks 0 and 48
Population: APTS included all randomized participants who received at least 1 dose of double-blind IMP. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lu AF82422
Number analyzed (Participants) | 28
ng/mL
  Week 0 | 5 (0)
  Week 48: number analyzed (Participants) | 23
  Week 48 | 1531 (886)

19. Secondary Outcome: Lu AF82422 CSF/Plasma Concentration Ratio in the DBP
Time Frame: Weeks 0 and 48
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lu AF82422
Number analyzed (Participants) | 28
ratio
  Week 0 | 25.00 (0.00)
  Week 48: number analyzed (Participants) | 23
  Week 48 | 0.40 (0.21)

ADVERSE EVENTS:
Time Frame: From date of first dose up to Week 88
Description: APTS included all randomized participants who received at least 1 dose of double-blind IMP.
Arm/Group | Placebo | Lu AF82422
All-Cause Mortality (participants affected / at risk) | 2/21 | 2/40
Serious Adverse Events (participants affected / at risk) | 7/21 | 12/40
Other Adverse Events (participants affected / at risk) | 14/21 | 34/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Lu AF82422 (N=40)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 2 (5)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Lu AF82422 (N=40)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 3 (3)
Injection site extravasation (General disorders) | 2 (2) | 1 (3)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 10 (10)
Urinary tract infection (Infections and infestations) | 2 (3) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3)
Blood triglycerides increased (Investigations) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 3 (3)
Low density lipoprotein increased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT05104476/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05104476/SAP_001.pdf